CLINICAL TRIAL: NCT02577705
Title: Building Wealth and Health Network: A Microfinance/TANF Demonstration Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Hunger-Free Communities (Other)
Responsible Party: Principal Investigator, Mariana Chilton, PhD, MPH, Principal Investigator, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1041002551
Record Dates: First submitted 2015-10-13; First posted 2015-10-16 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2015-10

CONDITIONS: Hunger; Child Development; Social Isolation
Keywords: food insecurity; adverse childhood experiences; violence exposure; trauma; poverty; TANF; assets; depression; randomized control trial
MeSH Terms: conditions — Social Isolation; Wounds and Injuries; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Self Empowerment Groups (Experimental): Intervention activities included helping participants to open savings accounts at a local federal credit union with 1:1 matches of up to twenty dollars per month for 12 months. Participants also received financial empowerment and Peer Support curriculum, weekly for about 3 hours per week for 28 weeks.
  Interventions: Behavioral: Self Empowerment Groups; Behavioral: Financial Empowerment; Behavioral: Matched Savings
- Financial Empowerment (Experimental): Intervention activities included helping participants to open savings accounts at a local federal credit union with 1:1 matches of up to twenty dollars per month for 12 months. Participants also received financial empowerment weekly for about 3 hours per week for 28 weeks.
  Interventions: Behavioral: Financial Empowerment; Behavioral: Matched Savings
- Control Group (No Intervention): The Control group did not receive assistance in opening a matched savings account, and were required by the County Assistance Office to participate in other Temporary Assistance for Needy Families (TANF) mandated work participation activities according to standard procedure.

INTERVENTIONS:
Behavioral: Self Empowerment Groups — The Self Empowerment Groups (SEG) curriculum draws key components from the S.E.L.F. tool within Sanctuary, focusing the four domains: creating personal, emotional, moral and physical safety (S), processing and managing emotions (E), recognizing loss and letting go (L), and developing goals for a sense of future (F). S.E.L.F. establishes a common language that all people who have experienced adversity can use to organize their lives and work towards building stable foundations to support their goals and invest in their potential.
  Arms: Self Empowerment Groups
Behavioral: Financial Empowerment — The Financial Empowerment curriculum developed for this study consisted of interactive exercises, worksheets, and journal assignments that fostered understanding and practice of banking, building credit and debt management, making the most of one's money, and setting financial goals for oneself and one's family. Content focused on identifying and harnessing the internal and external resources that participants can leverage to begin taking steps towards financial self-sufficiency.
  Arms: Financial Empowerment; Self Empowerment Groups
Behavioral: Matched Savings — Participants were assisted with opening a savings accounts at a local non-profit federal credit union (with 1:1 matches of up to twenty dollars per month) over the course of 12 months.
  Arms: Financial Empowerment; Self Empowerment Groups

SUMMARY:
The goals of the The Building Wealth and Health Network (The Network) are to develop and rigorously test an asset building model that will build financial, social and human capital through asset building, financial education and trauma-informed peer support. Program components include: 1) Matched savings accounts; 2) Financial literacy classes; and 3) Peer support groups using the Sanctuary ® trauma-informed approach to social services. This program is offered in partnership with the Department of Public Welfare of the Commonwealth of Pennsylvania. The program elements will fulfill work requirements for the program called temporary Assistance for Needy Families (TANF).

The hypothesis is that the program's combination of services will result in improved economic security through boosting income, increasing assets, and building a supportive social network, that then translates to better health outcomes.

DETAILED DESCRIPTION:
Families with young children under age six participating in The Temporary Assistance for NeedyFamilies Program (TANF) that are deemed "work mandatory" are required to participate in work-related activities for at least 20 hours per week in order to receive TANF benefits. However, due to financial hardship, poor health, and exposure to violence and adversity, the success families achieve through TANF participation can be limited.

In 2013, 45.3 million people lived in poverty in the United States, including over one in five children under the age of six, yet only 27% of eligible families received Temporary Assistance for Needy Families (TANF). While child poverty increases the risk of poor health and developmental delays, many public assistance programs, such as the Supplemental Nutrition Assistance Program (SNAP), the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC), and housing subsidies, protect vulnerable children from the negative effects of poverty. However, it is unclear if TANF has demonstrated significant improvements in maternal and child wellbeing, in moving families out of poverty, or in fully preparing low-income families for success in the workforce.

One of the goals of TANF is to provide job skills and education programs to support adults and their children as they enter the workforce. However, many families experience barriers to employment, which may prevent them from successfully transitioning off of TANF. This may be due in part to poor health among those receiving TANF, as approximately one third of TANF recipients have reported a work-limiting health condition; and almost 43% of TANF recipients reported multiple types of disability including memory impairment, emotional/mental limitations, movement limitations, and sensory impairment. In addition to the poor health and disability reported by TANF participants, they also report alarmingly high rates of exposure to violence and adversity in their communities and in their family relationships. For instance, among TANF eligible families, rates of intimate partner violence are as high as 74% compared to up to 31% in the general community, posing a major barrier to rates of employment. While exposure to violence in adulthood indicates severe hardship, such exposure to violence across the lifespan, reaching back into childhood, is also reported at significantly higher rates among low-income families. Adverse childhood experiences (ACEs) consisting of physical and emotional abuse and neglect, sexual abuse, and household dysfunction, such as having a household member in prison, or witnessing domestic violence are especially prevalent among those receiving TANF. ACEs and violence exposure are closely linked to work-limiting conditions such as depression, cardiovascular disease, food insecurity and other health conditions. Exposure to ACEs has been linked to higher rates of worker absenteeism and stress surrounding work and finances in adulthood, indicating an association between ACEs and later financial stability. Other related barriers to work are having a criminal record, or having served time in prison, and among female heads of household TANF recipients, the prevalence of interactions with the criminal justice system is quite high compared to other low income populations. Finally, when a parent of a young child is in prison, it can have detrimental effects on the child's development, which in turn, demands more attention, time and care by adult caregivers, creating more barriers to work. Female heads of households who have a criminal history are at greater risk for reaching the TANF time limit which can exacerbate the barriers of obtaining employment. Furthermore, children whose parents have a criminal history are at a greater risk of becoming involved in the criminal justice system and are more likely to exhibit high-risk behaviors than children in the general population.

The high levels of adversity among TANF recipients and those living in poverty is a significant concern because adversity impacts physical and mental health, academic achievement, employment, the development of executive skills such as working memory and cognitive controls, and parenting of the next generation. Emphasis on job search and work participation for families without attention to adversity and poor health can be a set up for failure. Preliminary evidence demonstrates that social support and comprehensive approaches to social work that build resilience may have strong success in limiting the negative impacts of exposure to violence and adversity. However, the majority of TANF programs across the country rarely integrate such approaches, and in many states, TANF participants that are unable to meet the mandated work requirements, potentially due to poor health and exposure to violence and adversity, may be more likely to be "sanctioned," either have their cash benefits reduced, or cut off completely for a duration of time.

Families that receive sanctions are more likely to have significant health barriers to work participation. Additionally, those that have been sanctioned reported higher rates of intimate partner violence, and physical and behavioral health problems. Sanctions can then increase hardships families already face. For instance, compared to families who have not been sanctioned, families that experience sanction report higher rates of household food insecurity, utility shut-offs, child hospitalizations, difficulty paying for health care, homelessness, and disruptions in children's schooling. This is especially problematic as those who are sanctioned often have young children, putting those children at increased risk during sensitive developmental phases.

To compound the mental and physical barriers to work and self-sufficiency, TANF-eligible families, like many low income families, have low financial literacy, poor no credit history, few or no assets, and are unbanked (having no checking or savings account) or under-banked (having a bank account, but still primarily relying on alternative financial services such as check cashing and money orders). In order to supplement meager income, families may resort to earning income and spending money through the informal economy where they are paying higher fees for check cashing, paying bills, and acquiring loans. This lack of access to mainstream financial institutions and activities can be crippling, as savings and other tangible assets play a critical role in helping shield families from unexpected income shocks, allowing families to weather periods of economic uncertainty without falling further into poverty. Savings create a financial foundation, increase economic security, and can be, over time, invested into education for children. Asset building activities show improvements in health, greater civic and community involvement, and lower rates in the intergenerational transfer of poverty. Savings can also reduce the extreme stress that often accompanies maternal depression. Finally, the positive impacts of savings have held true even during the recession.

In partnership with the state of Pennsylvania Health and Human Services Department, The Building Wealth and Health Network (The Network), a randomized, controlled pilot study, sought to evaluate effectiveness of an intervention to address family hardships associated with exposure to adversity and violence, social isolation, and low financial capability in order to help families get on the pathway to self-sufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of TANF cash benefits for four years or less, and
* Subject to mandatory TANF 20-hour work requirement, and
* Parents of at least one child below the age of six

Exclusion Criteria:

* Adults who are unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Change in family economic hardship | Quarterly change for up to 15 months
  Family economic hardship is a singular outcome captured in three measures of hardship:
  1) The U.S Household Food Security Survey Module (HFSSM) which measures food insecurity, 2) an energy security survey, which measures "energy insecurity," and 3) a housing security survey, which measures "housing instability." These three measures combine into a singular measure of hardship that consists of
  "No hardship" [no positive response to three hardships above] "Moderate hardship" [at least one of the three hardships] and "Severe hardship" [consisting of 2 or 3 hardships]

SECONDARY OUTCOMES:
Change in Career readiness | Quarterly change for up to 15 months
  Career readiness is measured using the employment hope scale.
Change in Mental Health | Quarterly change for up to 15 months
  To assess depressive symptoms among adult participants, we used the Center for Epidemiologic Studies Depression (CES-D).
Change in Child development | Quarterly change for up to 15 months
  Children's developmental status was measured by the Parents' Evaluations of Developmental Status Survey. Participants were asked ten questions about their child's developmental issues: global/cognitive, expressive language and articulation, fine-motor, gross motor, behavior, social-emotional, self-help, school, and any other concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Chilton, PhD, MPH, Principal Investigator — Drexel University
Locations (1):
- Drexel University School of Public Health, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Duncan GJ, Brooks-Gunn J. Family poverty, welfare reform, and child development. Child Dev. 2000 Jan-Feb;71(1):188-96. doi: 10.1111/1467-8624.00133. PMID 10836573
- [Background] Black MM, Quigg AM, Cook J, Casey PH, Cutts DB, Chilton M, Meyers A, Ettinger de Cuba S, Heeren T, Coleman S, Rose-Jacobs R, Frank DA. WIC participation and attenuation of stress-related child health risks of household food insecurity and caregiver depressive symptoms. Arch Pediatr Adolesc Med. 2012 May;166(5):444-51. doi: 10.1001/archpediatrics.2012.1. PMID 22566545
- [Background] Frank DA, Chilton M, Casey PH, Black MM, Cook JT, Cutts DB, Meyers AF. Nutritional-assistance programs play a critical role in reducing food insecurity. Pediatrics. 2010 May;125(5):e1267; author reply e1267-8. doi: 10.1542/peds.2010-0808. No abstract available. PMID 20435705
- [Background] Dworsky, A. and M.E. Courtney, Barriers to employment among TANF applicants and their consequences for self-sufficiency. Families in Society-the Journal of Contemporary Social Services, 2007. 88(3): p. 379-389.
- [Background] Trisi, D. and L. Pavetti, TANF Weakening as a Safety Net for Poor Families, in Center on Budget and Policy Priorities, http://www.cbpp.org/cms/index.cfm?fa=view&id=3700, Editor. 2012, Center on Budget and Policy Priorities: Washington, D.C
- [Background] Bloom, D., P.J. Loprest, and S.R. Zedlewski, TANf recipients with barriers to employment. Washington, DC: The Urban Institute. Temporary Assistance for Needy Families Program-Research Synthesis Brief, 2011. 1
- [Background] Loprest, P. and E. Maag, Disabilities among TANF recipients: Evidence from NHIS. 2009, The Urban Institute: Washington, D.C.
- [Background] Kennedy AC. Urban adolescent mothers exposed to community, family, and partner violence: prevalence, outcomes, and welfare policy implications. Am J Orthopsychiatry. 2006 Jan;76(1):44-54. doi: 10.1037/0002-9432.76.1.44. PMID 16569126
- [Background] Bowie, S.L. and D.M. Dopwell, Metastressors as barriers to self-sufficiency among TANF-reliant African American and Latina women. Affilia, 2013
- [Background] Lown EA, Schmidt LA, Wiley J. Interpersonal violence among women seeking welfare: unraveling lives. Am J Public Health. 2006 Aug;96(8):1409-15. doi: 10.2105/AJPH.2004.057786. Epub 2006 Jun 29. PMID 16809602
- [Background] Raphael J. Keeping battered women safe during welfare reform: new challenges. J Am Med Womens Assoc (1972). 2002 Winter;57(1):32-5. PMID 11905488
- [Background] Cheng TC. Intimate partner violence and welfare participation: a longitudinal causal analysis. J Interpers Violence. 2013 Mar;28(4):808-30. doi: 10.1177/0886260512455863. Epub 2012 Aug 27. PMID 22929347
- [Background] Adams AE, Bybee D, Tolman RM, Sullivan CM, Kennedy AC. Does job stability mediate the relationship between intimate partner violence and mental health among low-income women? Am J Orthopsychiatry. 2013 Oct;83(4):600-8. doi: 10.1111/ajop.12053. PMID 24164531
- [Background] Staggs SL, Long SM, Mason GE, Krishnan S, Riger S. Intimate partner violence, social support, and employment in the post-welfare reform era. J Interpers Violence. 2007 Mar;22(3):345-67. doi: 10.1177/0886260506295388. PMID 17308203
- [Background] Frogner, B., R. Moffit, and D. Ribar, Leaving Welfare: Long-Term Evidence from Three Cities. Baltimore, MD: Johns Hopkins University. https://orchid. hosts. jhmi. edu/wfp/files/WP10-01_Leaving% 20Welfare. pdf, 2010.
- [Background] Breiding MJ, Smith SG, Basile KC, Walters ML, Chen J, Merrick MT. Prevalence and characteristics of sexual violence, stalking, and intimate partner violence victimization--national intimate partner and sexual violence survey, United States, 2011. MMWR Surveill Summ. 2014 Sep 5;63(8):1-18. PMID 25188037
- [Background] Cambron C, Gringeri C, Vogel-Ferguson MB. Physical and mental health correlates of adverse childhood experiences among low-income women. Health Soc Work. 2014 Nov;39(4):221-9. doi: 10.1093/hsw/hlu029. PMID 25369722
- [Background] Danese A, Moffitt TE, Harrington H, Milne BJ, Polanczyk G, Pariante CM, Poulton R, Caspi A. Adverse childhood experiences and adult risk factors for age-related disease: depression, inflammation, and clustering of metabolic risk markers. Arch Pediatr Adolesc Med. 2009 Dec;163(12):1135-43. doi: 10.1001/archpediatrics.2009.214. PMID 19996051
- [Background] Anda RF, Brown DW, Dube SR, Bremner JD, Felitti VJ, Giles WH. Adverse childhood experiences and chronic obstructive pulmonary disease in adults. Am J Prev Med. 2008 May;34(5):396-403. doi: 10.1016/j.amepre.2008.02.002. PMID 18407006
- [Background] Ross CE, Mirowsky J. Neighborhood disadvantage, disorder, and health. J Health Soc Behav. 2001 Sep;42(3):258-76. PMID 11668773
- [Background] Chilton M, Knowles M, Rabinowich J, Arnold KT. The relationship between childhood adversity and food insecurity: 'It's like a bird nesting in your head'. Public Health Nutr. 2015 Oct;18(14):2643-53. doi: 10.1017/S1368980014003036. Epub 2015 Jan 22. PMID 25611561
- [Background] Anda RF, Fleisher VI, Felitti VJ, Edwards VJ, Whitfield CL, Dube SR, Williamson DF. Childhood Abuse, Household Dysfunction, and Indicators of Impaired Adult Worker Performance. Perm J. 2004 Winter;8(1):30-8. doi: 10.7812/TPP/03-089. PMID 26704603
- [Background] Phillips, S.D. and A.J. Dettlaff, More than parents in prison: The broader overlap between the criminal justice and child welfare systems. Journal of Public Child Welfare, 2009. 3(1): p. 3-22.
- [Background] Travis, J., Families and Children of Offenders Who Return Home. Fed. Probation, 2005. 69: p. 31
- [Background] Head, V.B., C.E., Ovwigho, P, Criminal History as an employment barrier for TANF recipients. 2009, University of Maryland Baltimore: Baltimore.
- [Background] Lu W, Mueser KT, Rosenberg SD, Jankowski MK. Correlates of adverse childhood experiences among adults with severe mood disorders. Psychiatr Serv. 2008 Sep;59(9):1018-26. doi: 10.1176/ps.2008.59.9.1018. PMID 18757595
- [Background] Evans, G.W., J. Brooks-Gunn, and P.K. Klebanov, Stressing out the poor: Chronic physiological stress and the income-achievement gap. Community Investments, 2011(Fall): p. 22-27.
- [Background] Liu Y, Croft JB, Chapman DP, Perry GS, Greenlund KJ, Zhao G, Edwards VJ. Relationship between adverse childhood experiences and unemployment among adults from five U.S. states. Soc Psychiatry Psychiatr Epidemiol. 2013 Mar;48(3):357-69. doi: 10.1007/s00127-012-0554-1. Epub 2012 Aug 7. PMID 22869349
- [Background] Farah MJ, Shera DM, Savage JH, Betancourt L, Giannetta JM, Brodsky NL, Malmud EK, Hurt H. Childhood poverty: specific associations with neurocognitive development. Brain Res. 2006 Sep 19;1110(1):166-74. doi: 10.1016/j.brainres.2006.06.072. Epub 2006 Aug 1. PMID 16879809
- [Background] Noble KG, McCandliss BD, Farah MJ. Socioeconomic gradients predict individual differences in neurocognitive abilities. Dev Sci. 2007 Jul;10(4):464-80. doi: 10.1111/j.1467-7687.2007.00600.x. PMID 17552936
- [Background] Randles, J.M., Partnering and Parenting in Poverty: A Qualitative Analysis of a Relationship Skills Program for Low-Income, Unmarried Families. Journal of Policy Analysis and Management, 2014. 33(2): p. 385-412.
- [Background] Larkin H, Felitti VJ, Anda RF. Social work and adverse childhood experiences research: implications for practice and health policy. Soc Work Public Health. 2014;29(1):1-16. doi: 10.1080/19371918.2011.619433. PMID 24188292
- [Background] Larkin H, MacFarland NS. Restorative integral support (RIS) for older adults experiencing co-occurring disorders. Int J Aging Hum Dev. 2012;74(3):231-41. doi: 10.2190/AG.74.3.d. PMID 22844693
- [Background] Pavetti, L., M.K. Derr, and H. Hesketh, Review of sanction policies and research studies. report from Mathematica Policy Research, Inc., to the Office of the Assistant Secretary for Planning and Evaluation, US Department of Health and Human Services (March 2003), 2003.
- [Background] Lindhorst T, Mancoske RJ. The Social and Economic Impact of Sanctions and Time Limits on Recipients of Temporary Assistance to Needy Families. J Sociol Soc Welf. 2006 Mar;33(1):93-114. PMID 18080002
- [Background] Lens, V., Work sanctions under welfare reform: Are they helping women achieve self-sufficiency. Duke J. Gender L. & Pol'y, 2006. 13: p. 255
- [Background] Pavetti, L., et al., The use of TANF work-oriented sanctions in Illinois, New Jersey, and South Carolina. Washington, DC: Mathematica Policy Research, Inc, 2004
- [Background] Cook JT, Frank DA, Berkowitz C, Black MM, Casey PH, Cutts DB, Meyers AF, Zaldivar N, Skalicky A, Levenson S, Heeren T. Welfare reform and the health of young children: a sentinel survey in 6 US cities. Arch Pediatr Adolesc Med. 2002 Jul;156(7):678-84. doi: 10.1001/archpedi.156.7.678. PMID 12090835
- [Background] Kalil, A., K.S. Seefeldt, and H.c. Wang, Sanctions and material hardship under TANF. Social Service Review, 2002. 76(4): p. 642-662.
- [Background] Oggins, J. and A. Fleming, Welfare reform sanctions and financial strain in a food-pantry sample. J. Soc. & Soc. Welfare, 2001. 28: p. 101
- [Background] Reichman, N.E., J.O. Teitler, and M.A. Curtis, TANF Sanctioning and Hardship. The Social Service Review, 2005. 79(2): p. 215-236,403-404.
- [Background] Larson, A.M., S. Singh, and C. Lewis, Sanctions and Education Outcomes for Children in TANF Families. Child & Youth Services, 2011. 32(3): p. 180-199.
- [Background] Stegman, M.A. and R. Faris, Welfare, work and banking: The use of consumer credit by current and former TANF recipients in Charlotte, North Carolina. Journal of Urban Affairs, 2005. 27(4): p. 379-402.
- [Background] Zhan, M., S.G. Anderson, and J. Scott, Financial management knowledge of the low-income population: Characteristics and needs. Journal of Social Service Research, 2006. 33(1): p. 93-106
- [Background] Anderson, S., M. Zhan, and J. Scott, Improving the knowledge and attitudes of low-income families about banking and predatory financial practices. Families in Society: The Journal of Contemporary Social Services, 2007. 88(3): p. 443-452.
- [Background] Sullivan, J.X., Welfare Reform, Saving, and Vehicle Ownership Do Asset Limits and Vehicle Exemptions Matter? Journal of human resources, 2006. 41(1): p. 72-105.
- [Background] FDIC Unbanked/Underbanked Survey Study Group, 2011 FDIC National Survey of Unbanked and Underbanked Households, F.D.E. Corportaion, Editor. 2012, Federal Deposit Ensurance Corportaion: Washington, D.C.
- [Background] Sherraden, M.W., Assets and the poor: a new American welfare policy. 1991, Armonk, N.Y.: M.E. Sharpe. xviii, 324 p.
- [Background] Shapiro, T.M. and E.N. Wolff, Assets for the poor: the benefits of spreading asset ownership. The Ford Foundation series on asset building. 2001, New York: Russell Sage Foundation. xiv, 389 p.
- [Background] Sherraden, M.W., Inclusion in the American dream: assets, poverty, and public policy. 2005, New York: Oxford University Press. xxii, 409 p.
- [Background] Shanks, T.R. and C. Robinson, Over-stressed kids: Examining the impact of economic security on children and families, A.E. Casey, Editor. 2011: Baltimore, MD.
- [Background] Brooks, J. and K. Wiedrich, Assets & Opportunity Scorecard: A Portrait of financial insecurity and Policies to Rebuild Prosperity in America, in CFED, http://scorecard.cfed.org, Editor. 2012: Washington, D.C.
- [Background] Hendey, L., S.-M. McKernan, and B. Woo, Weathering the Recession: The Financial Crisis and Family Wealth Changes in Low-Income Neighborhoods, T.A.E.C.F.a.t.U. Institute, Editor. 2012: Baltimore, MD, and Washington, DC.
- [Background] Hong, P., J. Polanin, and T. Pigott, Validation of the Employment Hope Scale: measuring psychological self-sufficiency among low-income jobseekers. Research on Social Work Practice, 2012. 22(3): p. 323-332.
- [Background] Hong, P.Y.P., The employment hope scale: Measuring an empowerment pathway to employment success. 2013, Loyola University Chicago
- [Background] Schwarzer, R., Jerusalem, M., Generalized Self-Efficacy scale, in Measures in health psychology: A user's portfolio. Causal and control beliefs, J. Weinman, Wright, S., Johnston, M., Editor. 1995, NFER-NELSON: Windsor, England. p. 35-37.
- [Background] Bickel, G., et al., Guide to measuring household food security. US Department of Agriculture, Food and Nutrition Service, Office of Analysis, Nutrition, and Evaluation. http://www. fns. usda. gov/fsec/FILES/Guide% 20to% 20Measuring% 20Household% 20Food% 20Security (3-23-00). pdf, 2000.
- [Background] Bickel, G., et al., Measuring Food Security in the United States: Guide to Measuring Household Food Security. 2000, US Department of Agriculture, Food and Nutrition Service, Office of Analysis and Evaluation: Alexandria, VA.
- [Background] Cook JT, Frank DA, Casey PH, Rose-Jacobs R, Black MM, Chilton M, Ettinger de Cuba S, Appugliese D, Coleman S, Heeren T, Berkowitz C, Cutts DB. A brief indicator of household energy security: associations with food security, child health, and child development in US infants and toddlers. Pediatrics. 2008 Oct;122(4):e867-75. doi: 10.1542/peds.2008-0286. PMID 18829785
- [Background] Cutts DB, Meyers AF, Black MM, Casey PH, Chilton M, Cook JT, Geppert J, Ettinger de Cuba S, Heeren T, Coleman S, Rose-Jacobs R, Frank DA. US Housing insecurity and the health of very young children. Am J Public Health. 2011 Aug;101(8):1508-14. doi: 10.2105/AJPH.2011.300139. Epub 2011 Jun 16. PMID 21680929
- [Background] Blake, K.S., R.L. Kellerson, and A. Simic, Measuring overcrowding in housing. Washington, DC: Department of Housing and Urban Development, Office of Policy Development and Research, 2007.
- [Background] Casey P, Goolsby S, Berkowitz C, Frank D, Cook J, Cutts D, Black MM, Zaldivar N, Levenson S, Heeren T, Meyers A; Children's Sentinel Nutritional Assessment Program Study Group. Maternal depression, changing public assistance, food security, and child health status. Pediatrics. 2004 Feb;113(2):298-304. doi: 10.1542/peds.113.2.298. PMID 14754941
- [Background] Radloff, L.S., The CES-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1977. 1: p. 385-401
- [Background] Hann D, Winter K, Jacobsen P. Measurement of depressive symptoms in cancer patients: evaluation of the Center for Epidemiological Studies Depression Scale (CES-D). J Psychosom Res. 1999 May;46(5):437-43. doi: 10.1016/s0022-3999(99)00004-5. PMID 10404478
- [Background] Zhang W, O'Brien N, Forrest JI, Salters KA, Patterson TL, Montaner JS, Hogg RS, Lima VD. Validating a shortened depression scale (10 item CES-D) among HIV-positive people in British Columbia, Canada. PLoS One. 2012;7(7):e40793. doi: 10.1371/journal.pone.0040793. Epub 2012 Jul 19. PMID 22829885
- [Background] Glascoe, F.P., Scoring, Administration and Interpretation Guidelines, in Collaborating with parents: Using Parents' Evaluation of Developmental Status to detect and address developmental and behavioral problems. 1998, Ellsworth & Vandermeer Press: Nashville, TN, US. p. 9-30.
- [Background] Glascoe FP. Using parents' concerns to detect and address developmental and behavioral problems. J Soc Pediatr Nurs. 1999 Jan-Mar;4(1):24-35. doi: 10.1111/j.1744-6155.1999.tb00077.x. PMID 10334009
- [Background] Dong M, Anda RF, Felitti VJ, Dube SR, Williamson DF, Thompson TJ, Loo CM, Giles WH. The interrelatedness of multiple forms of childhood abuse, neglect, and household dysfunction. Child Abuse Negl. 2004 Jul;28(7):771-84. doi: 10.1016/j.chiabu.2004.01.008. PMID 15261471
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Richters, J.E. and W. Saltzman, Survey of Exposure to Community Violence: Parent report version. 1990: J.E. Richters.
- [Background] Scarpa, A., et al., Community Violence Exposure in University Students A Replication and Extension. Journal of Interpersonal Violence, 2002. 17(3): p. 253-272.
- [Background] Osborne, C. and J. Knab, Work, welfare, and young children's health and behavior in the Fragile Families and Child Wellbeing Study. Children and Youth Services Review, 2007. 29(6): p. 762-781.
- [Background] Wildeman, C., Paternal Incarceration and Children's Physically Aggressive Behaviors Evidence from the Fragile Families and Child Wellbeing Study. Social Forces, 2010. 89(1): p. 285-309.
- [Background] Schwarzer, R., Everything you wanted to know about the General Self-Efficacy Scale but were afraid to ask: documentation of the General Self-Efficacy Scale. 2014.
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219
- [Derived] Sun J, Patel F, Kirzner R, Newton-Famous N, Owens C, Welles SL, Chilton M. The Building Wealth and Health Network: methods and baseline characteristics from a randomized controlled trial for families with young children participating in temporary assistance for needy families (TANF). BMC Public Health. 2016 Jul 16;16:583. doi: 10.1186/s12889-016-3233-4. PMID 27421287